CLINICAL TRIAL: NCT04522544
Title: A Phase II Study of Immunotherapy With Durvalumab (MEDI4736) and Tremelimumab in Combination With Y-90 SIRT for Intermediate Stage HCC
Brief Title: Durvalumab and Tremelimumab in Combination With Y-90 SIRT for Intermediate Stage HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: AstraZeneca (Industry); Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMMUWIN; 2019-004597-26 (EudraCT Number); ESR-19-14400 (Other Grant/Funding Number: AstraZeneca); AIO-HEP-0319/ass (Other: AIO-Studien-gGmbH); IKF027 (Other: IKF Trial ID); 2024-513950-32-00 (EU CTIS Number)
Record Dates: First submitted 2020-08-04; First posted 2020-08-21 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma Non-resectable; HCC
Keywords: hepatocellular carcinoma; intermediate stage HCC; SIRT; Durvalumab; Tremelimumab; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIRT (Arm A) (Experimental): Y-90 SIRT + Tremelimumab + Durvalumab
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Procedure: Y-90 SIRT
- TACE (Arm B) (Experimental): DEB-TACE + Tremelimumab + Durvalumab
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Procedure: DEB-TACE

INTERVENTIONS:
Drug: Tremelimumab — 300 mg Tremelimumab C1D1
Drug: Durvalumab — 1500 mg Durvalumab C1D1 + Q4W (max. 13 cycles)
Procedure: Y-90 SIRT — Locoregional therapy will be performed as a standard-of-care procedure
  Arms: SIRT (Arm A)
Procedure: DEB-TACE — Locoregional therapy will be performed as a standard-of-care procedure
  Arms: TACE (Arm B)

SUMMARY:
A Phase II study of immunotherapy with Durvalumab (MEDI4736) and Tremelimumab in combination with Y-90 SIRT for intermediate stage HCC

DETAILED DESCRIPTION:
The IMMUWIN phase II will test the safety and anti-tumor efficacy of the combination of Durvalumab and Tremelimumab with Y-90 SIRT.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
2. Age ≥ 18 years at time of study entry.
3. Body weight > 30 kg.
4. Multinodular or large, solitary HCC, not eligible for resection or local ablation.
5. Histologically confirmed diagnosis of HCC.
6. Scheduled to receive locoregional therapy as standard of care.
7. At least one measurable site of disease as defined by RECIST 1.1criteria with spiral CT scan or MRI.
8. No prior systemic anti-cancer therapy.
9. Child-Pugh A.
10. Performance status (PS) ≤ 1 (ECOG scale).
11. Life expectancy of at least 12 weeks.
12. Adequate blood count, liver-enzymes, and renal function:

    * Hemoglobin ≥ 9.0 g/dL, absolute neutrophil count ANC ≥1.5 (or 1.0) x (> 1500 per mm^3), platelets ≥100 (or 75) x 10^9/L (>75,000 per mm^3);
    * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN);
    * AST (SGOT), ALT (SGPT) ≤ 2.5 x institutional ULN unless liver metastases are present, in which case it must be ≤5x ULN;
    * International normalized ratio (INR) ≤ 1.25.
13. Albumin ≥ 31 g/dL.
14. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
15. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial and must use two effective forms of contraception if sexually active.
16. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving IMP and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational products (Durvalumab and Tremelimumab). Women who are not of childbearing potential (i.e. who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception).
17. If patient has concurrent Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection, meets the following criteria:

    * Patients with HBV or HCV infection should be monitored for viral levels during study participation;
    * Patients with detectable hepatitis B surface antigen (HBsAg) or detectable HBV DNA should have HBV DNA < 100 IU/ml and should be managed per local treatment guidelines. Controlled (treated) hepatitis B subjects will be allowed if they started treatment at the time point of enrollment into the study by the latest and treatment is continued during study participation and for ≥ 6 months after end of study treatment;
    * HCV patients with advanced HCC are mostly not treated for their HCV infection. However, patients treated for HCV are considered suitable for inclusion if antiviral therapy has been completed prior to first administration of study drug.
18. Subject is willing and able to comply with the protocol for the duration of the study including

Exclusion Criteria:

1. Diffuse HCC or presence of vascular invasion or extrahepatic spread with the following exception:

   o Invasion of a segmental portal vein or hepatic veins.
2. Patients with advanced liver disease as defined below:

   o liver cirrhosis with stage Child Pugh B and C.
3. Any contraindications for hepatic embolization procedures:

   * Known hepatofugal blood flow;
   * Known porto-systemic shunt;
   * Impaired clotting test (platelet count < 70 x 10^9/L, INR > 1.25);
   * Renal failure/insufficiency requiring hemo-or peritoneal dialysis;
   * Known severe atheromatosis;
   * Total thrombosis or total invasion of the main branch of the portal vein.
4. Locoregional therapies ongoing or completed < 4 weeks prior to the baseline scan.
5. History of cardiac disease:

   * Congestive heart failure > New York Heart Association (NYHA) class 2;
   * Active coronary artery disease (CAD) (myocardial infarction ≥ 6 months prior to study entry is allowed);
   * Cardiac arrhythmias (Grade > 2 NCI-CTCAE Version 5.0) which are poorly controlled with anti-arrhythmic therapy or requiring pace maker;
   * Uncontrolled hypertension;
   * Clinically significant gastrointestinal bleeding within 4 weeks prior to start of study drug.
6. Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months prior to the first dose of study drug with the exception of thrombosis of a segmental portal vein.
7. Prior, systemic anti-cancer therapy, radiotherapy administered < 4 weeks prior to study entry, endocrine- or immunotherapy or use of other investigational agents.
8. Current or prior use of immunosuppressive medication within 14 days before the first dose of Durvalumab or Tremelimumab. The following are exceptions to this criterion:

   * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
   * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
   * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
9. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
10. Major surgery within 4 weeks of starting the study and patients must have recovered from effects of major surgery.
11. Patients with second primary cancer, except adequately treated basal skin cancer or carcinoma in-situ of the cervix, unless curatively treated and disease-free for 3 years or longer.
12. Any co-existing medical condition that in the investigator's judgement will substantially increase the risk associated with the patient's participation in the study.
13. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
14. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
15. History of allogenic organ transplantation.
16. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or compliance with the study protocol.
17. Symptomatic brain metastases. A scan to confirm the absence of brain metastases is required in the presence of corresponding symptoms.
18. Pregnant or breast-feeding women.
19. Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
20. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
21. Known allergy or hypersensitivity to any of the IMPs or any of the constituents of the product.
22. Is currently participating or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
23. Patient who has been incarcerated or involuntarily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) [according to RECIST 1.1] at 6 months. | 6 months
  Proportion of allocated subjects with best response of complete or partial response

SECONDARY OUTCOMES:
Progression free survival (PFS) | Time from the date of randomization to the date of first observed disease progression or death (approx. 42 months)
  Time from the date of randomization to the date of first observed disease progression (investigator assessment according to RECIST 1.1) or death from any cause.
Overall survival (OS) | From the date of treatment Date of enrollment until date of death if applicable (up to 42 months until Study Closure)
  Overall survival will be determined as time from the date of treatment allocation to the date of death.
Treatment related SAEs | From first patient included until study closure (approx. 42 months after First Patient Included)
  Treatment related serious adverse events rate (SAE) will be determined. All observed toxicities and side effects will be graded according to NCI CTCAE v5.0 for all patients and the degree of association of each with the study treatment assessed and summarized.
Overall response rate (ORR) as best overall response (BOR) during therapy | 13 months
  ORR as BOR during therapy will be defined as the proportion of allocated subjects with best response of complete or partial response from date of randomization until disease progression or death from any cause occurs.
Overall response rate (ORR) at 6 months | 6 months
  ORR at 6 months for patients who received single treatment of TACE/SIRT
Quality of Life (QoL) | 24 months
  Quality of life will be assessed by the European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC QLQ-C30 questionnaire) and will be evaluated based on the EORTC QLQ-C30 scoring manual in its most current version at time of data analysis.

OTHER OUTCOMES:
Translational research | 3 months
  Exploratory: Correlation analysis between selected molecular parameters and clinical data to identify molecular biomarkers predictive for outcome are not fully defined at the time this protocol is written. The optional translational research program will consider the latest research data available at the time of analysis. Analysis might comprise (but is not limited to) staining for PD-L1 protein expression on tumor cells using the commercially available IVD Kits (22C3 pharmDx assay, DAKO North America) and lymphocytes, testing for expression of PD-1, PD-L1 and PD-L2, Immune cell infiltrates (IGHM, CD3, CD8, FOXP3, CD68, CD205), Chemokines (CXCL9. CXCL10, CXCL13) and invasion markers (MMP7, MMP9) and assessing circulating nucleic acids and tumor specific transcripts.

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Director — Frankfurter Institut für Klinische Krebsforschung IKF GmbH; Arndt Vogel, Prof. Dr., Principal Investigator — Hannover Medical School
Locations (12):
- Germany (12):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Universtitätsklinikum Schleswig-Holstein, Lübeck
  - Klinikum rechts der Isar der Technischen Universität München, München
  - München Klinik Bogenhausen, München
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.